CLINICAL TRIAL: NCT07330375
Title: The Effect of Intravenous Combination Dexmedetomidine - Ketamine Versus Dexmedetomidine on Post-Operative Analgesia in Patients Undergoing Vaginal Hysterectomy Under Spinal Anesthesia
Brief Title: Effect of Intravenous Dexmedetomidine and Ketamine on Post-Operative Analgesia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, abdelrahman elsayed abdelrahman elsayed saad amer, Resident of Anesthesia, Intensive Care and Pain management, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1088
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Analgesia; Postoperative Pain Management
Keywords: spinal anesthesia; vaginal hysterectomy; dexmedetomidine; ketamine
MeSH Terms: interventions — Dexmedetomidine; Ketamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either group Dexmedetomidine-ketamine combination (receiving I/V of dexmedetomidine 0.5 µg/kg over 10 min ,followed by 0.5 µg/kg/hr infusion and receiving I/V of ketamine 0.2mg/kg over 2-3min ,followed by 0.2 mg/kg/hr infusion ) OR group Dexmedetomidine (receiving I/V of dexmedetomidine 0.5 µg/kg over 10 min ,followed by 0.5 µg/kg/hr infusion and receiving I/V of normal saline ) through sequentially numbered opaque sealed envelope. Anesthesiologist and patients both will be blinded to the administered drug in two groups. Either of the drugs will be injected after giving spinal anesthesia and confirmation of achievement of desired level of block.
  In both groups, Dexmedetomidine will titrate by 0.1 µg/kg/h every 30 min to maintain a Ramsay Sedation Scale (RSS) score of 3-4. If the RSS score was >4 at 0.2 µg/kg/h of Dexmedetomidine, both drug infusions were stopped.The drug infusions were restarted at the lowest doses at RSS of 3.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the drugs will be prepared by anesthesiologist who will not be the part of the study and these drugs will be injected by another anesthesiologist who will be blinded to the drugs and will be participating into the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group D+K (Dexmedetomidine-Ketamine Combination) (Active Comparator): Patients will receive intravenous dexmedetomidine (drug 1) loading dose of 0.5 µg/kg diluted with normal saline to a volume of 10 ml solution over 10 min (started when a sensory level of T10 was achieved) Maintenance dose of 0.5 µg/kg/h infusion and Intravenous ketamine (drug 2) loading dose of 0.2mg/kg diluted with normal saline to a volume of 10 ml solution over 2-3min ( started when a sensory level of T10 was achieved) maintenance dose of 0.2 mg/kg/h infusion.
  In both groups, drug 1 will be titrated by 0.1 µg/kg/h every 30 min to maintain a Ramsay Sedation Scale (RSS) score of 3-4.
  If the RSS score was >4 at 0.2 µg/kg/h of Drug 1, both drug infusions will be stopped.The drug infusions will be restarted at the lowest doses at RSS of 3.
  Interventions: Drug: Dexmedetomidine; Drug: Ketamine
- Dexmedetomidine group (D) (Placebo Comparator): Patients will receive intravenous dexmedetomidine (drug 1) loading dose of 0.5 µg/kg diluted with normal saline to a volume of10 ml solution over 10 min (started when a sensory level of T10 was achieved) Maintenance dose of 0.5 µg/kg/h and intravenous normal saline (drug 2) loading dose 10ml of solution over 2-3min ( started when a sensory level of T10 was achieved) and a maintenance dose of 0.2 mg/kg/h as placebo.
  In both groups, drug 1 will be titrated by 0.1 µg/kg/h every 30 min to maintain a Ramsay Sedation Scale (RSS) score of 3-4. If the RSS score >4 at 0.2 µg/kg/h of Drug 1, both drug infusions will be stopped.The drug infusions will be restarted at the lowest doses at RSS of 3.
  Interventions: Drug: Dexmedetomidine; Drug: Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous dexmedetomidine 0.5 µg/kg diluted with normal saline to a volume of 10 ml solution over 10 min followed by 0.5 µg/kg/h infusion.
Drug: Ketamine — Intravenous ketamine 0.2 mg/kg diluted with normal saline to a volume of 10 ml solution over 2-3 min followed by 0.2 mg/kg/hr infusion.
  Arms: Group D+K (Dexmedetomidine-Ketamine Combination)
Drug: Saline (0.9% NaCl) — intravenous normal saline 10ml of solution over 2-3min followed by 0.2 mg/kg/hr infusion as placebo
  Arms: Dexmedetomidine group (D)

SUMMARY:
In this study the participants aim to Compare The Effect of Intravenous Combination Dexmedetomidine _ Ketamine versus Dexmedetomidine on Post-Operative Analgesia In Vaginal Hysterectomy Proceeded Under Spinal Anesthesia regarding efficacy, hamemodynamic stability, outcomes and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will accept written informed consent.
* Age: 21-65 years old.
* Sex: female.
* BMI: <35 kg/m2
* Physical status: American Society of Anesthesiology (ASA) of Grade I-II
* Type of operation: vaginal hysterectomy under spinal anesthesia.

Exclusion Criteria:

* Uncooperative patients
* Any contraindication for spinal anesthesia e.g. coagulopathy, infection at site of block, and hypersensitivity to any drug used in this study.
* Patients who are known to be drug dependent.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female aged b/w 21-65 years
Enrollment: 50 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Assess the postoperative analgesic requirements in first 24 hours. | Pain grade of patients will be evaluated immediately on arrival to PACU then at 2, 4, 6,12, 24 hours postoperatively
  Pain will be assessed and recorded using visual analogue scale (VAS) {0=no pain, 1 to 3 = mild pain, 4 to 6 = moderate pain, 7 to 10 = severe pain} immediately on arrival to PACU then at 2, 4, 6,12, 24 hours after surgery by an observer blinded to treatment groups. • On the first analgesic demand or when VAS scale 1-3, diclofenac 75 mg IV will be given. nalbupine 20 mg IV will be administered as a rescue analgesic, as needed if the VAS scale 4-10 .

SECONDARY OUTCOMES:
Total amount of rescue analgesic requirement | In first 24 hours postoperatively
  Total amount of rescue analgesic requirement in first 24 hours Postoperatively

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Result] Pandya MJ, Shah A. Comparative evaluation of dexmedetomidine and ketamine for epidural analgesia in lower limb orthopedic surgeries [Internet]. Indian J Clin Anaesth. 2020 [cited 2025 Dec 29];7(1):166-171. Available from: https://doi.org/10.18231/j.ijca.2020.029
- [Result] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Result] Moawad NS, Santamaria Flores E, Le-Wendling L, Sumner MT, Enneking FK. Total Laparoscopic Hysterectomy Under Regional Anesthesia. Obstet Gynecol. 2018 Jun;131(6):1008-1010. doi: 10.1097/AOG.0000000000002618. PMID 29742667
- [Result] DOI: 10.33545/26643766.2021.v4.i3a.280
- [Result] DOI: 10.9734/jpri/2022/v34i43A36310
- [Result] Krishna AS, Agarwal J, Khanuja S, Kumar S, Khan A, Butt KM. Comparison of intravenous dexmedetomidine versus ketamine-dexmedetomidine combination on spinal block characteristics in patients undergoing lower limb orthopaedic surgery - A randomised clinical trial. Indian J Anaesth. 2024 Sep;68(9):795-800. doi: 10.4103/ija.ija_14_24. Epub 2024 Aug 16. PMID 39386403
- [Result] Blaudszun G, Lysakowski C, Elia N, Tramer MR. Effect of perioperative systemic alpha2 agonists on postoperative morphine consumption and pain intensity: systematic review and meta-analysis of randomized controlled trials. Anesthesiology. 2012 Jun;116(6):1312-22. doi: 10.1097/ALN.0b013e31825681cb. PMID 22546966